CLINICAL TRIAL: NCT00015821
Title: A Pilot Study of Thalidomide as an Inhibitor of Angiogenesis in the Treatment of Myelofibrosis With Myeloid Metaplasia (MMM)
Brief Title: Thalidomide in Treating Patients With Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01853; NCI-2012-01853 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000068367; NCCTG-N9982; N9982 (Other: North Central Cancer Treatment Group); N9982 (Other: CTEP); U10CA025224 (NIH)
Record Dates: First submitted 2001-05-06; First posted 2003-05-23 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Primary Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — Thalidomide

ARMS (1):
- Treatment (thalidomide) (Experimental): Patients receive oral thalidomide once daily for 1 year in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease may receive 1 additional year of therapy.
  Interventions: Drug: thalidomide; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: thalidomide — Given PO
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of thalidomide in treating patients who have myelofibrosis. Thalidomide may stop the growth of myelofibrosis by stopping blood flow to the cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate whether thalidomide, a potent inhibitor of angiogenic and fibrogenic growth factors, is an effective therapeutic agent in patients with MMM. Specifically, to assess whether thalidomide improves anemia and/or organomegaly in patients with MMM.

II. To assess the effects of thalidomide on the myelofibrotic stroma with respect to microvascular architecture and angiogenesis, collagen and reticulin deposition, and the expression of the mediating growth factors bFGF, TGF-b, and PDGF, and their respective receptors.

OUTLINE: This is a multicenter study.

Patients receive oral thalidomide once daily for 1 year in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease may receive 1 additional year of therapy.

Patients are followed every 6 months until 5 years from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed myelofibrosis with myeloid metaplasia

  * Agnogenic myeloid metaplasia
  * Post-polycythemic myeloid metaplasia
  * Post-thrombocythemic myeloid metaplasia
* No metastatic carcinoma, lymphoma, myelodysplasia, hairy cell leukemia, mast cell disease, acute leukemia (including M7), or acute myelofibrosis
* No chromosomal translocation t(9;22) or bcr/abl gene rearrangement
* Presence of reticulin fibrosis in bone marrow and leukoerythroblastosis and dacrocytosis in peripheral blood
* Presence of anemia (hemoglobin less than 10 g/dL), palpable splenomegaly, or hepatomegaly
* Performance status - ECOG 0-2
* Absolute neutrophil count greater than 750/mm^3
* Platelet count less than 400,000/mm^3
* WBC less than 50,000/mm^3
* Bilirubin no greater than 2 mg/dL (if total bilirubin elevated, direct bilirubin must be normal)
* AST no greater than 3 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 3 times ULN
* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile women must use at least 1 highly active method AND 1 additional effective method of contraception for at least 4 weeks before study, during study, and for at least 4 weeks after study
* Fertile men must use effective contraception during study and for at least 4 weeks after study
* No uncontrolled infection
* No concurrent condition that would preclude study
* No peripheral neuropathy
* At least 1 month since prior interferon, pirfenidone, anagrelide, or epoetin alfa
* At least 1 month since prior hydroxyurea or other chemotherapy
* At least 1 month since prior corticosteroids or androgen derivatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2000-05; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Confirmed Response, i.e., an objective status of complete or partial response, recorded on 2 consecutive evaluations at least 4 weeks apart. | Up to 5 years
  The proportion of successes will be estimated using the Binomial point estimator (number of successes divided by the total number of evaluable patients) and 95% confidence intervals calculated using the Duffy-Santner algorithm for multi-stage designs.

SECONDARY OUTCOMES:
Survival | Number of days from registration date to the date of death or last follow-up, assessed up to 5 years
  Kaplan-Meier survival curves will be generated to estimate survival.
Time to progression | Number of days from registration date to the date of disease progression or last follow-up, assessed up to 5 years
  Kaplan-Meier survival curves will be generated to estimate time to progression.
Response duration | Number of days from the first date that objective status = complete or partial response was recorded to the date of disease progression or date of death, whichever comes first, assessed up to 5 years
  Kaplan-Meier survival curves will be generated to estimate response duration.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Elliott, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States